CLINICAL TRIAL: NCT02999321
Title: The Effects of Aspartame on Appetite, Body Composition and Oral Glucose Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Ajinomoto USA, INC. (Industry)
Responsible Party: Principal Investigator, Richard Mattes, Professor of Nutrition Sciences, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 055-045
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Oral Glucose Tolerance
MeSH Terms: interventions — Aspartame; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0% aspartame (water) (Experimental): participants will not have any aspartame, this is a control.
  Interventions: Other: water
- 5 mg aspartame (Experimental): participants will receive 5 mg aspartame in a beverage.
  Interventions: Other: aspartame
- 15mg aspartame (Experimental): participants will receive 5 mg aspartame in a beverage, and 10mg in capsules.
  Interventions: Other: aspartame

INTERVENTIONS:
Other: aspartame — will be given 5mg aspartame or 15 mg aspartame
  Arms: 15mg aspartame; 5 mg aspartame
Other: water — control group
  Arms: 0% aspartame (water)

SUMMARY:
Assess the impact of chronic use of aspartame on glycemia, appetite and body composition.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of three parallel arms: 0% (water), 5 mg, 15mg aspartame. Participants will have an oral glucose tolerance test at the beginning and end of a 12 week intervention. . Participants will report to the lab weekly for 12 weeks to pick up their next week's intervention products and measurements for body weight, waist circumference, blood pressure and heart rate. They will consume their intervention products daily for 12 weeks. They will record appetite sensations and collect a 24 hour urine sample at weeks 0, 4, 8, and 12.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25
* Fasting blood sugar between 72 and 108 mg/dl via capillary finger-stick.

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
change oral glucose tolerance | week 0 4 hours
  sample taken at time point 0
change oral glucose tolerance | week 0 4 hours
  sample taken at time point 15 minutes post glucola
change oral glucose tolerance | week 0 4 hours
  sample taken at time point 30 minutes post glucola
change oral glucose tolerance | week 0 4 hours
  sample taken at time point 60 minutes post glucola
change oral glucose tolerance | week 0 4 hours
  sample taken at time point 90 minutes post glucola
change oral glucose tolerance | week 0 4 hours
  sample taken at time point 120 minutes post glucola
change oral glucose tolerance | week 0 4 hours
  sample taken at time point 180 minutes post glucola
change oral glucose tolerance | week 0 4 hours
  sample taken at time point 240 minutes post glucola
change oral glucose tolerance | week 12 4 hours
  sample taken at time point 0
change oral glucose tolerance | week 12 4 hours
  sample taken at time point 15 minutes post glucola
change oral glucose tolerance | week 12 4 hours
  sample taken at time point 30 minutes post glucola
change oral glucose tolerance | week 12 4 hours
  sample taken at time point 60 minutes post glucola
change oral glucose tolerance | week 12 4 hours
  sample taken at time point 90 minutes post glucola
change oral glucose tolerance | week 12 4 hours
  sample taken at time point 120 minutes post glucola
change oral glucose tolerance | week 12 4 hours
  sample taken at time point 180 minutes post glucola
change oral glucose tolerance | week 12 4 hours
  sample taken at time point 240 minutes post glucola

SECONDARY OUTCOMES:
Appetite | every hour for 1 day at week 0
  questionnaire on hunger, fullness, desire to eat, prospective consumption, thirst taken hourly for one day.
Appetite | every hour for 1 day at week 4
  questionnaire on hunger, fullness, desire to eat, prospective consumption, thirst taken hourly for one day
Appetite | every hour for 1 day at week 8
  questionnaire on hunger, fullness, desire to eat, prospective consumption, thirst taken hourly for one day
Appetite | every hour for 1 day at week 12
  questionnaire on hunger, fullness, desire to eat, prospective consumption, thirst taken hourly for one day
Body composition | week 0
  body composition measurement Plysmography (BOD POD)
Body composition | week 12
  body composition measurement Plysmography (BOD POD)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue Univeristy, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Higgins KA, Considine RV, Mattes RD. Aspartame Consumption for 12 Weeks Does Not Affect Glycemia, Appetite, or Body Weight of Healthy, Lean Adults in a Randomized Controlled Trial. J Nutr. 2018 Apr 1;148(4):650-657. doi: 10.1093/jn/nxy021. PMID 29659969